CLINICAL TRIAL: NCT06282874
Title: An Open-label, Single-arm, Multicenter, Prospective Study of Lorlatinib in Patients With ALK-Positive NSCLC With Brain or Leptomeningeal Metastases
Brief Title: Lorlatinib in Patients With ALK-Positive NSCLC With Brain or Leptomeningeal Metastases
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2303
Record Dates: First submitted 2024-01-30; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Brain Metastases; Leptomeningeal Metastasis
Keywords: ALK-Positive Non-Small-Cell Lung Cancer; Brain Metastases; Leptomeningeal Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Meningeal Carcinomatosis | interventions — lorlatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BM/LM cohort (Experimental): Fifty eligible subjects will be divided into a BM cohort (brain parenchymal metastasis only) and an LM cohort (leptomeningeal metastasis ± brain parenchymal metastasis)
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib 100 mg once daily on days 1 to 28 of each 28-day cycle
  Other Names: PF-06463922

SUMMARY:
This study is an investigator-initiated, prospective, open-label, single-arm, multicenter clinical trial aimed at exploring the antitumor activity of Lorlatinib in ALK-positive NSCLC patients with brain/ leptomeningeal metastases.

DETAILED DESCRIPTION:
Fifty eligible subjects will be divided into a BM cohort (brain parenchymal metastasis only) and an LM cohort (leptomeningeal metastasis ± brain parenchymal metastasis). All subjects will receive Lorlatinib 100 mg once daily on days 1 to 28 of each 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender not restricted.
2. Histologically or cytologically confirmed NSCLC patients.
3. ALK rearrangement positive confirmed by FISH, RT-PCR, IHC Ventana D5F3 or NGS. Patients with other treatable gene mutations besides ALK need to submit for discussion with the study experts to determine eligibility.
4. Patients who are treatment-naive or have undergone treatment are both eligible for enrollment. If the first-line treatment prior to the trial was an ALK inhibitor or chemotherapy, there must be a washout period of at least 28 days before the first trial drug administration. In case of disease worsening, the study experts can be consulted to decide if the washout period can be shortened.
5. Adverse Events related to the previous systemic treatment must have recovered to ≤ grade 1 (CTCAE 5.0) or to pre-treatment levels, except for AEs that the investigator does not consider to pose a safety risk to the patient.
6. At least one CNS lesion that meets the following criteria: 1. Imaging and/or cerebrospinal fluid suggestive of leptomeningeal metastasis. Imaging-identified leptomeningeal metastasis does not require cerebrospinal fluid confirmation; 2. Brain metastasis confirmed by Magnetic Resonance Imaging (MRI), with ≥3 brain lesions; or 1-2 lesions that are unsuitable for surgical treatment or the patient refuses surgical treatment. For patients without leptomeningeal metastasis, there must be at least one measurable lesion with a diameter of ≥5mm in the brain.
7. Patients with or without brain/leptomeningeal metastasis-related symptoms are eligible.
8. The subject's expected survival time must be 12 weeks or longer.
9. For patients without leptomeningeal metastasis, Eastern Cooperative Oncology Group Performance (ECOG) score of 0-2; for patients with leptomeningeal metastasis, ECOG score of 0-3.
10. Participants must have normal primary organ function.
11. For women of childbearing potential (defined as not being postmenopausal for at least 1 year, or having undergone surgical sterilization or hysterectomy), a serum pregnancy test should be conducted within seven days prior to the first administration of the investigational drug, and the result should be negative. All participants (regardless of gender) must agree to use contraceptive measures during the entire treatment period and for at least 90 days after the last dose of the investigational drug.

Participants must understand and voluntarily sign the written informed consent form, demonstrate good compliance, adhere to the trial treatment plan and visit schedule, and be able to cooperate in observing adverse events and treatment efficacy.

Exclusion Criteria:

1. Have received treatment with the investigational drug or known allergy to the ingredients or excipients of the investigational drug.
2. Concurrent participation in another clinical study, except for observational (non-interventional) clinical studies or subsequent stages of interventional studies, excluding patients who have received treatment with any other investigational drug within 28 days before the start of the study treatment.
3. Brain metastasis with bleeding, or the presence of central nervous system complications requiring urgent local intervention (such as surgery, radiotherapy, etc.).
4. Presence of spinal cord compression unless pain symptoms and neurological function have remained stable or improved 2 weeks prior to enrollment.
5. Received open surgery (except surgery for biopsy purposes) within ≤14 days prior to enrollment.
6. Fever with a temperature above 38℃ within the past week; or clinically significant bacterial, fungal or viral infection, including but not limited to HIV infection, active HCV infection, active tuberculosis; or infections requiring hospitalization, septicemia, severe pneumonia, etc.
7. Significant clinical abnormalities in rhythm, conduction, or morphology on resting ECG, such as complete left bundle branch block, 2nd degree or higher heart block, clinically significant ventricular arrhythmia or atrial fibrillation.
8. Unstable angina, congestive heart failure (NYHA class III or IV), myocardial infarction, coronary/peripheral artery bypass, cerebrovascular accident, untreated transient ischemic attack, or symptomatic pulmonary embolism occurring currently or within the past 3 months.
9. Past or current clinically active interstitial lung disease; current radiation pneumonia requiring corticosteroid treatment.
10. Disorders of swallowing function, active gastrointestinal disease, or other diseases significantly affecting the absorption, distribution, metabolism, and excretion of the investigational drug. History of major gastric resection.
11. Presence of other acquired, congenital immunodeficiency diseases, or previous solid organ or hematopoietic stem cell transplantation.
12. Evidence of severe or uncontrolled systemic diseases (such as severe mental, neurological diseases, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension i.e., still being greater than or equal to CTCAE 5.0 grade 3 hypertension after drug treatment).
13. Use or consumption of known potent CYP3A4 inhibitors in medications or food within the past 2 weeks; use of known potent CYP3A4 inducers within the past 2 weeks; use of medications that act as CYP3A4 substrates (with a narrow therapeutic index) within the past 2 weeks.
14. Severe acute or chronic mental illness, including recent (within the past year) or active suicidal ideation or behavior.
15. For pregnant or lactating women or male or female participants with reproductive potential, refusal to adopt effective contraceptive measures during the treatment period and for 90 days after the last use of the investigational drug.
16. The investigator believes that the participant may be unable to complete the study or comply with the study requirements.
17. The investigator believes that there are other potential risks making the participant unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
intracranial objective response rate（iORR） | From date of the first dose of lorlatinib treatment until the date of last follow up or death, up to 18 months.
  BM Cohort: percentage of participants demonstrating an intracranial complete response or partial response according to modified RECIST v1.1 criteria; LM Cohort: percentage of participants demonstrating an intracranial complete response or partial response according to the imaging criteria of RANO-LM.

SECONDARY OUTCOMES:
Progression-free survival (PFS) and intracranial PFS（iPFS） | From date of the first dose of lorlatinib treatment until the date of last follow up or death, up to 18 months.
  PFS defined as time from the first dose of lorlatinib to the first documentation of progression or death from any cause. Specifically, intracranial PFS pertains to the progression of the disease confined within the brain.
Obiective response rate (ORR) | From date of the first dose of lorlatinib treatment until the date of last follow up or death, up to 18 months.
  ORR defined as assessed percentage of participants demonstrating a complete response or partial response including central nervous system disease, extracranial disease and overall disease.
Disease control rate (DCR) and intracranial disease control rate (iDCR) | From date of the first dose of lorlatinib treatment until the date of last follow up or death, up to 18 months.
  Disease Control Rate, is determined by assessing the percentage of participants who achieve a best response of confirmed Complete Response (CR), confirmed Partial Response (PR), or exhibit stable disease for various disease sites including central nervous system, extracranial, and leptomeningeal involvement, as well as overall disease status. Specifically, intracranial DCR focuses on evaluating the disease control rate within the brain.
Overall survival | From date of the first dose of lorlatinib treatment until the date of last follow up or death, up to 18 months.
  Overall survival defined as time from the start of treatment until death or last follow-up
Number of participants with adverse events | From date of the first dose of lorlatinib treatment until the date of last follow up or death, up to 18 months.
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ji Yang, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial Perople's Hospital, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No